CLINICAL TRIAL: NCT06624709
Title: The Benefit in Terms of Improvement in Haemoglobin Level at 6 Months in Premature Babies Receiving Alternate Iron Substitution 4 Times a Week Compared to a Daily Substitution
Acronym: BienFER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riccardo Pfister (Other)
Responsible Party: Sponsor-Investigator, Riccardo Pfister, Head of neonatology department, Principal Investigator, Clinical Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-02374
Record Dates: First submitted 2024-09-14; First posted 2024-10-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-10

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alternate (4 times/week) iron supplementation (Active Comparator): This arm will receive 2-3mg/kg/d of maltofer 4 times a day
  Interventions: Drug: Iron Supplement
- Daily iron substitution (Sham Comparator): This arm will receive 2-3mg/kg/d of maltofer 7 times per week.
  Interventions: Drug: Iron Supplement

INTERVENTIONS:
Drug: Iron Supplement — The interventional group will receive 2-3mg/kg/day of iron supplementation 4 times per week and the sham comparator will receive 2-3mg/kg/day of iron supplementation 7 times per week

SUMMARY:
BienFer is a double-blinded randomized controlled trial about iron substitution and abdominal pain. Premature babies and low birth weight babies have lower iron stores than term newborns and are therefore at greater risk of iron deficiency and anemia. Iron deficiency could have consequences for cerebral development. Ferric substitution reduces the risk of iron deficiency and anemia. It is common to replace premature babies with iron substitution between 2 weeks and 6 months of life. In practice, the medical staff notice that newborn with iron substitution have abdominal pain and constipation. A study in the adult population shows that alternate iron supplementation versus daily supplementation improved iron absorption, with no difference in hemoglobin level and decrease abdominal pain. Studies in children shows that intermittent iron supplementation do not change hemoglobin and ferritin level and improve adherence. There is no data comparing daily versus alternate supplementation in premature babies.

The aim of the study is to evaluate if alternate (4 times/week) iron supplementation is equivalent to daily iron substitution for hemoglobin values in premature babies between 28 0/7 weeks amenorrhea (WA) and 34 6/7 WA, and if it reduces abdominal discomfort and inflammation, and if it improves compliance.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies between 28 0/7WA and 34 6/7 WA
* Parental consent, postnatal
* Age of 2 weeks

Exclusion Criteria:

* anemia < 80g/l at 2 weeks of age
* Intraventricular Hemorrhage stage III and IV
* Necrotizing Enterocolitis
* Enteral feeding less than 100ml/kg/j after 2 weeks of life
* Congenital disorder

Ages: 14 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Anemia at 6 months | 6 months
  Hemoglobin level

SECONDARY OUTCOMES:
Anemia | at 2weeks, 1 month, 2-3 months
  Hemoglobin
Anemia | at 2weeks, 1 month, 2-3 months
  Hematocrit level
Ferritin | at 2 weeks, 1 month, 2-3 months and 6 months
  Ferritin
Ret-Hb level | at 2 weeks, 1 month, 2-3 months and 6 months
  Ret-Hb level
Transfusion | at 1 month, 2-3 months and 6 months
  Number of patients needed a transfusion
Therapeutic level | at 1 month, 2-3 months and 6 months
  Number of patients needed to increase the iron substitution to a therapeutic level
Evaluation of abdominal inflammation | at 2 weeks and 2-3 months
  Calprotectin level
Evaluation of abdominal inflammation | at 2 weeks and 2-3 months
  Hepcidin level
Evaluation of intestinal microbiota | at 2-3 months
  Fecal sequencing
Comorbidities | at 6 months
  Number of retinopathy of prematurity (ROP)
Comorbidities | at 6 months
  Number of periventricular leukomalacia (PVL)
Comorbidities | at 6 months
  Number of sepsis
Comorbidities | at 6 months
  Number of intraventricular hemorrhage (IVH)
Comorbidities | at 6 months
  Number of bronchopulmonary dysplasia (BPD)
Comorbidities | at 6 months
  Number of necrotizing enterocolitis (NEC)
Evaluation of weight gain | at 2 weeks, 1 month, 2-3 months and 6 months
  Tracking weight in Kilograms
Evaluation of height gain | at 2 weeks, 1 month, 2-3 months and 6 months
  Tracking height in Centimeters
Evaluation of the growth's parameter | at 2 weeks, 1 month, 2-3 months and 6 months
  Tracking head circumference in Centimeters
Evaluation of abdominal discomfort | 3 times per week during hospitalization then 1 time per 2 weeks until 6 months
  Edin scale (0 (better outcome, no pain)-15 (worse outcome, pain))
Evaluation of abdominal discomfort | 3 times per day during hospitalization then 1 time per 2 weeks until 6 months
  Classify stools with Bristol scale (1 (severe constipation) -7 (severe diarrhea))

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - HUG, Geneva, Canton of Geneva
  - CHUV, Lausanne, Canton of Vaud